CLINICAL TRIAL: NCT06835907
Title: Investigating the Efficacy of Baclofen in Patients with Alcohol Use Disorder (AUD) and Comorbid Anxiety Symptoms
Brief Title: Baclofen for Anxiety and Alcohol Use Disorder (AUD): an Open Label Study
Acronym: BAC2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1432024000205
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Alcohol use disorder (AUD); Baclofen; Anxiety
MeSH Terms: conditions — Alcoholism; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Baclofen (Experimental): SIngle arm study, investigating baclofen as standard care uptitrated to maximal tolerated dosage upon clinical judgment and not part of the trial. The active intervention involves questionnaires.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires include: the Alcohol Use Disorder Identification Test (AUDIT), Composite Autonomic Symptom Score (COMPASS-31), Depression Anxiety Stress Scale (DASS-21), Drug Desire Questionnaire (DDQ), Drinking Motives Questionnaire short form (DMQ-SF), Mini International Neuropsychiatric Interview (MINI), PROMIS-alcohol, Timeline Follow Back (TLFB) and Visual Analog Scale for craving (VAS).

SUMMARY:
The goal of this clinical trial is to determine the efficacy of baclofen for the treatment of alcohol use disorder (AUD) in patients with or without comorbid anxiety symptoms. The main questions it aims to answer are:

* Do we see more abstinent days after the study period in patients with high anxiety symptoms compared to low anxiety symptoms?
* Do we observe additional differences between patients with high- and low anxiety symptoms in: any drinking at the end of treatment (yes/no), number of patients who respond to treatment, anxiety score reduction, autonomic responses, craving scores, drinking motives and side effects?

Participants already taking baclofen as part of routine clinical care for treatment of AUD will be asked to answer several questionnaires over a 6 week study period.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-5 criteria for AUD
* Able to understand and provide written consent
* Already receiving baclofen or started with baclofen at start of hospitalization
* Therapeutic desire towards alcohol abstinence

Exclusion Criteria:

* Concurrent substance use disorder other than nicotine or cannabis
* Clinically significant psychiatric illness that requires pharmacotherapy, unless stable and no changes in medication has been made in the last 30 days
* Clinically significant medical diseases that may pose a risk to continuing baclofen use
* Pregnant or currently breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of days abstinent | Weekly during 6 week study period
  Number of days abstinent during baclofen treatment between AUD patients with and without comorbid anxiety, as measured by the TLFB.

SECONDARY OUTCOMES:
Any drinking | After 6 week study period
  Any drinking (i.e. drinking yes or no at the end of treatment) between AUD patients with and without comorbid anxiety, as measured by the TLFB.
Treatment response | After 6 week study period
  Number of individuals who respond to baclofen treatment, defined as reducing their alcohol use by more than 30% over the 6 week study period, as measured by the TLFB.
Autonomic symptom responses | At start and after 6 week study period
  Autonomic symptom responses measured by the COMPASS-31 assessing 6 domains of autonomic symptoms: orthostatic intolerance, vasomotor, secretomotor, gastro-intestinal, bladder and pupillomotor.
Craving scores | Weekly for the VAS and bi-weekly for the DDQ during the 6 week study period
  Craving scores measured by self-report VAS for craving and the DDQ.
Anxiety score reduction | At start and after 6 week study period
  Reduction in anxiety score measured using the DASS-21.
Drinking motives | At start of 6 week study period
  Drinking motives measured using the DMQ-SF.
Side effects | Weekly during 6 week study period
  Side effects assessed by open end questions

CONTACTS AND LOCATIONS:
Overall Officials: Cleo L Crunelle, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided